CLINICAL TRIAL: NCT07001189
Title: Impact of Regional Anesthesia on Inflammatory Mechanisms During Vaso-occlusive Crisis in Sickle Cell Patients
Acronym: ALRCVO-MP
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de la Guadeloupe (Other)
Responsible Party: Sponsor
Other Study IDs: PAP_RIPH3_2024/02; 2024-A00950-47 (Other: ANSM Frech Human Health Organisation)
Record Dates: First submitted 2025-05-23; First posted 2025-06-03 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Sickle Cell; Sickle Cell Disease; Vaso-Occlusive Crises
Keywords: Loco-regional anesthesia; inflammation; Vaso-Occlusive Crises
MeSH Terms: conditions — Anemia, Sickle Cell; Vaso-Occlusive Crises; Inflammation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Collection of two blood tubes for the quantification of protein and cytokine levels, and for the quantitative and qualitative analysis of circulating blood microparticles.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- RA-Group: When a sickle cell patient comes to the emergency department with pain such as vaso-occlusive crises, we will offer them the opportunity to participate in the study. Inclusion will therefore occur before the choice of analgesic technique. The patient will receive the treatment they have chosen (with or without regional anesthesia). Depending on their choice and/or any contraindications (e.g., morphine intolerance or allergy to ropivacaine), they will be placed in the "RA group" (if they received regional anesthesia) or the "non-RA group" (if they did not receive it).
- Non-RA group: When a sickle cell patient comes to the emergency department with pain such as vaso-occlusive crises, we will offer them the opportunity to participate in the study. Inclusion will therefore occur before the choice of analgesic technique. The patient will receive the treatment they have chosen (with or without regional anesthesia). Depending on their choice and/or any contraindications (e.g., morphine intolerance or allergy to ropivacaine), they will be placed in the "RA group" (if they received regional anesthesia) or the "non-RA group" (if they did not receive it).

SUMMARY:
Sickle cell disease is a chronic disease characterized by multiple vaso-occlusive complications. The basic treatment for patients with a vaso-occlusive crisis (VOC) is based on adequate hydration, oxygen therapy and pain control. Loco Regional Anesthesia (LRA) is one of the major treatments in resuscitation anesthesia for both anesthesia and analgesia. LRA allows effective and almost immediate pain control by blocking nerve afferents in a given area. LRA could decrease the inflammatory response during crises and accelerate resolution of the crisis.

DETAILED DESCRIPTION:
Regional anesthesia (RA) possesses intrinsic anti-inflammatory properties and can modulate the inflammatory response. For instance, ropivacaine reduces inflammation induced in vitro in rat epithelial cells. At the cellular level, lidocaine decreases free radical production by neutrophils, inhibits leukocyte phagocytic activity, and significantly suppresses cytokine production in response to endotoxemia.

The value of RA no longer lies solely in its ability to block nociceptive input via sodium channel inhibition. A peripheral nerve block with local anesthetics inhibits local neurogenic inflammation, thereby reducing sensitization, hyperalgesia, and the risk of pain chronification. A peripheral nerve block is therefore an anti-inflammatory treatment.

However, no study has yet demonstrated the anti-inflammatory effects of RA at the cellular level in sickle cell disease patients.

The aim of this study is to analyze the evolution of inflammatory markers during vaso-occlusive crises (e.g., MPs, cytokines, NETs, etc.), by comparing patients who received RA to those who did not during hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* patients adult >18 years
* patients with vaso-occlusive crisis

Exclusion Criteria:

* Pregnant or breastfeeding women
* Blood transfusion within the last 3 months
* Lack of affiliation with the French social security system
* Protected individuals

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult sickle cell patients consulting for vaso-occlusive crisis in CHU de Guadeloupe
Sampling Method: Non-Probability Sample
Enrollment: 34 (Estimated)
Dates: Start 2025-02-05 (Actual); Primary Completion 2027-02-05 (Estimated); Study Completion 2027-02-05 (Estimated)

PRIMARY OUTCOMES:
Inflammatory process during vaso-occlusive crises | Baseline and Day 1
  The variation between D0 and D1 in the proportion of endothelial cells expressing ICAM-1 on their surface, following stimulation with microparticles from patients who received or did not receive regional anesthesia.

SECONDARY OUTCOMES:
Quantification of protein levels | Baseline and day 1
  ICAM-1, VCAM-1, P-selectin, Elastase (marker of neutrophil extracellular traps (NET)
Quantification of cytokine levels | Baseline and day 1
  Quantification of cytokine levels
Quantitative and qualitative profil of blood microparticles | Baseline and day 1
  Quantitative and qualitative profil of blood microparticles

CONTACTS AND LOCATIONS:
Overall Officials: Amelie Rolle, MD, Principal Investigator — CHU de la Guadeloupe
Locations (1):
- Chu de La Guadeloupe, Pointe-à-Pitre, Guadeloupe

IPD SHARING:
Plan to Share IPD: Undecided